CLINICAL TRIAL: NCT00629759
Title: Phase 1 Clinical Study for Evaluating the Safety and Efficacy of a Transdermal Injection of JX-594 (Thymidine Kinase (-)/GM-CSF(+) Vaccinia Virus) Within the Tumor of Patients With Hepatic Carcinoma
Brief Title: A Study of Recombinant Vaccinia Virus to Evaluate the Safety and Efficacy of a Transdermal Injection Within the Tumor of Patients With Primary or Metastatic Hepatic Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jennerex Biotherapeutics (Industry)
Collaborators: Green Cross Corporation (Industry)
Responsible Party: David Kirn, MD, President and CEO, Jennerex, Inc. (Jennerex Biotherapeutics)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JX594-IT-HEP001
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2008-02

CONDITIONS: Neoplasms, Liver
Keywords: Jennerex; unresectable liver tumors; primary liver cancer; metastatic liver cancer; oncolytic virus; vaccinia virus; Pexa-Vec
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Vaccinia | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 1e8 pfu (plaque forming units)total dose each treatment day
  Interventions: Genetic: JX-594: Recombinant vaccinia virus (TK-deletion plus GM-CSF)
- 2 (Experimental): 3e8 pfu (plaque forming units) total dose each treatment day
  Interventions: Genetic: JX-594: Recombinant vaccinia virus (TK-deletion plus GM-CSF)
- 3 (Experimental): 1e9 pfu (plaque forming units) total dose each treatment day
  Interventions: Genetic: JX-594: Recombinant vaccinia virus (TK-deletion plus GM-CSF)
- 4 (Experimental): 3e9 pfu (plaque forming units) total dose each treatment day
  Interventions: Genetic: JX-594: Recombinant vaccinia virus (TK-deletion plus GM-CSF)

INTERVENTIONS:
Genetic: JX-594: Recombinant vaccinia virus (TK-deletion plus GM-CSF) — The total dose is divided between 1-3 tumors located within the liver. Patients are treated with JX-594 once every 3 weeks until progression at the site(s) of injection or until the patient has received a maximum of 4 treatments.

SUMMARY:
The primary purpose of this study is to determine the maximum tolerable dose (MTD) and/or the maximum feasible dose (MFD), as well as to evaluate the safety of JX-594 (Pexa-Vec) injected within hepatic carcinoma tumors.

DETAILED DESCRIPTION:
Patients are treated with JX-594 once every three weeks until progression at the site(s) of injection or until the patient has received a maximum of 4 treatments; four additional cycles can be administered to patients with an objective response of the injected tumor(s) (i.e. 8 total treatments possible). Study dose levels are 1e8 pfu, 3e8 pfu, 1e9 pfu and 3e9 pfu per treatment. Standard Phase I dose-escalation guidelines are used, with 2-6 patients enrolled per cohort (3 if no dose-limiting toxicities are reported).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with hepatic carcinoma (primary or metastatic) clinically or histologically confirmed to have tumors (≤10cm maximum diameter) that are progressing (refractory to standard treatment) despite regular treatment and that can be transdermally accessed by an injection needle in an imaging-guided procedure
* Tumor progression despite undergoing regular treatment such as surgery, transarterial chemoembolization, chemotherapy, and radiotherapy
* Performance score: Karnofsky Performance Score (KPS) ≥70
* Expected survival of at least 16 weeks
* For patients who are sexually active, able and willing to use contraceptives for a three month period during and after taking JX-594
* WBC > 3,500 cells/mm3
* ANC > 1,500 cells/mm3
* Hemoglobin > 10g/dL
* Platelet count > 75,000 plts/mm3
* Serum creatinine < 1.5 mg/dL
* AST, ALT < 2.5 x ULN
* Total bilirubin ≤ 2.0 mg/dL
* In patients with primary HCC, Child Pugh A or B
* Able/willing to sign an IRB/IEC/REB-approved written consent form
* Able and willing to comply with study procedures and follow-up examinations

Exclusion Criteria:

* Pregnant or nursing an infant
* Known infection with HIV
* Clinically significant active infection or uncontrolled medical condition considered high risk for investigational new drug treatment
* Significant immunodeficiency due to underlying illness (e.g. hematological malignancies, congenital immunodeficiencies and/or HIV infection/AIDS) and/or medication (e.g. high-dose systemic corticosteroids)
* Patients with household contacts with significant immunodeficiency
* History of exfoliative skin condition (e.g. severe eczema, ectopic dermatitis, or similar skin disorder) that at some stage has required systemic therapy
* Severe or unstable cardiac disease
* Use of adrenal cortical hormone drug or immunosuppressant within four weeks of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerable dose (MTD) and/or the maximum feasible dose (MFD), as well as to evaluate the safety of JX-594 injected within unresectable solid tumor(s) within the liver | Safety evaluation throughout study participation

SECONDARY OUTCOMES:
Secondary objectives include determination of JX-594 pharmacokinetics, replication and shedding, immune response, and injection site tumor responses.

CONTACTS AND LOCATIONS:
Overall Officials: David Kirn, MD, Study Director — Jennerex Biotherapeutics (Jennerex, Inc.)
Locations (1):
- Dong-A University Hospital, Busan, South Korea

REFERENCES:
- [Derived] Park BH, Hwang T, Liu TC, Sze DY, Kim JS, Kwon HC, Oh SY, Han SY, Yoon JH, Hong SH, Moon A, Speth K, Park C, Ahn YJ, Daneshmand M, Rhee BG, Pinedo HM, Bell JC, Kirn DH. Use of a targeted oncolytic poxvirus, JX-594, in patients with refractory primary or metastatic liver cancer: a phase I trial. Lancet Oncol. 2008 Jun;9(6):533-42. doi: 10.1016/S1470-2045(08)70107-4. Epub 2008 May 19. PMID 18495536
- See also: Sponsor company website — http://www.jennerex.com